CLINICAL TRIAL: NCT03019692
Title: Longterm Outcome of Children With Neonatal Intra-Ventricular or Intra-Cranial Hemorrhage (IVH, ICH)
Brief Title: Longterm Outcome of Children With Neonatal Intra-Ventricular or Intra-Cranial Hemorrhage
Acronym: NEONATAL ICH
Status: Recruiting | Type: Observational
Sponsor: Laniado Hospital (Other)
Responsible Party: Principal Investigator, Laniado Hospital, Liana.Adani, Laniado Hospital
Other Study IDs: 0148-16-LND-2016121
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Neonates Premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- enrolled babies with neonatal intracranial bleed: all babies who suffered from intra cranial or intraventricular bleed during neonatal period

SUMMARY:
Intraventricular hemorrhage (IVH) is the most commonly recognized cerebral lesion on ultrasound in extremely preterm infants. Papile classification is commonly used to grade the severity of IVH. Grade III-IV IVH and other lesions noted on ultrasound including periventricular leukomalacia (pvl) porencephaly, and ventriculomegaly are well Documented to be associated with adverse neurodevelopmental outcomes.

However, the true impact of lower-grade IVH on the neurodevelopment of these extreme preterm infants has not been well described.

Also Neurodevelopmental outcome for neonatal non-traumatic Intra Cranial Hemorrhage (ICH) is not well established.

The aim of this study is to look retrospectively at babies with neonatal IVH or ICH and follow their radiological, cognitive, motor and functional outcomes.

The study will focus on postnatal files, and on images performed as part of the child's follow-up during hospitalization and after discharge.

DETAILED DESCRIPTION:
The study will be performed as a Retrospective chart review with key words : IVH, ICH of babies discharged from Laniado Hospital Neonatal care service or ICU, or being followed in the pediatric neurosurgical clinic and prematurity/neonatology clinic of the hospital.

All charts of such children will be included, to review clinical, and radiological available data.

Registration of Clinical, Radiological data as presented or submitted by the parents on Neurosurgical neonatology and Neurological Followups will be performed by PI or CI and coded in the data anonymously.

Follow up will be performed as clinically indicated without addition of any specific studies due to the research.

The endpoints of the study:

primary endpoint:

1. How many children needed surgical intervention related to the hemorrhage (ICH, IVH) secondary endpoints:
2. Clinical and functional outcome of children - REGARDING normal schooling, need for assistance in ADL in difference from the parallel normal child.

correlation between the type of hemorrhage, clinical data related to gestational age and weight at birth, and outcomes will be performed.

ELIGIBILITY:
Inclusion Criteria:

newborns or premature babies who suffered intra-cranial or intra-ventricular hemorrhage children who are followed by PI in the neurosurgical clinic in Laniado hospital and suffered from ICH or IVH and were treated elsewhere after birth -

Exclusion Criteria:

loss to followup within the first year after birth

-

Ages: 1 Hour to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: newborns or premature babies who suffered intra-cranial or intra-ventricular hemorrhage within the first 3 months after birth or before discharge after delivery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
need for surgery related to neonatal hemorrhage | 3 years

SECONDARY OUTCOMES:
normal schooling according to age | 6 years
need for ADL assistance beyond acceptable per age | 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sharon Nechama, Laniado Hospital, Netanya, Israel, Israel